CLINICAL TRIAL: NCT03631706
Title: An Adaptive Phase III, Multicenter, Randomized, Open-Label, Controlled Study of M7824 (Bintrafusp Alfa) Versus Pembrolizumab as a First-line Treatment in Patients With PD-L1 Expressing Advanced Non-small Cell Lung Cancer
Brief Title: M7824 Versus Pembrolizumab as a First-line (1L) Treatment in Participants With Programmed Death-ligand 1 (PD-L1) Expressing Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0037; 2018-001517-32 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: M7824; Pembrolizumab; PD-L1-tumor Expression; INTR@PID Lung 037; Bintrafusp alfa
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- M7824 (Experimental)
  Interventions: Drug: M7824
- Pembrolizumab (Active Comparator)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: M7824 — Participants received intravenous infusion of M7824 at a dose of 1200 milligrams (mg) once every 2 weeks until confirmed progression of disease, death, unacceptable toxicity, or study withdrawal.
  Arms: M7824
Drug: Pembrolizumab — Pembrolizumab: Participants received intravenous infusion of Pembrolizumab at a dose of 200 milligrams (mg) once every 3 weeks until confirmed progression of disease, death, unacceptable toxicity, or study withdrawal.
  Arms: Pembrolizumab

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bintrafusp alfa (M7824) compared with pembrolizumab in participants with advanced NSCLC with high PD-L1-tumor expression, with no epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) translocation. The Phase III adaptive design allows for the option to recruit up to 584 patients based on pre-specified rules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced NSCLC
* Have not received prior systemic therapy treatment for their advanced/Stage four NSCLC. Completion of treatment with cytotoxic chemotherapy, biological therapy, and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease. Confirmation of resolution of toxic effects of previous neoadjuvant/adjuvant chemotherapy therapy to Grade less than or equal to 1. For radiation toxicity or prior major surgeries, participants should have recovered from side effects and/or complications
* Have measurable disease based on RECIST 1.1
* Have a life expectancy of at least 3 months
* Availability of tumor tissue (less than 6 months old) before the first dose is mandatory to determine PD-L1 expression level prior to enrollment
* PD-L1 high status as determined by central testing
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with nonsquamous NSCLC histologies whose tumor harbors any of the following molecular alterations and targeted therapy is locally approved: epidermal growth factor receptor (EGFR) sensitizing (activating) mutation, anaplastic lymphoma kinase (ALK) translocation, ROS1 rearrangement, or BRAF V600E mutation
* Has received major surgery within 4 weeks prior to the first dose of study intervention; received thoracic radiation therapy of greater than 30 units of gray (Gy) within 6 months prior to the first dose of study
* Known severe hypersensitivity to investigational products (M7824 or pembrolizumab), or any components in their formulations
* Previous malignant disease (other than the target malignancy to be investigated in this study) within the last 3 years
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (119):
- United States (25):
  - Oncology Specialties, PC; Clearview Cancer Institute, Huntsville, Alabama
  - Cedars Sinai Medical Center - Inflammatory Bowel Disease Center (Clinic, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Kaiser Permanente - Harbor City, San Diego, California
  - Sansum Clinic - Santa Barbara, Santa Barbara, California
  - Rocky Mountain Cancer Centers - Colorado Springs, N. Nevada, Colorado Springs, Colorado
  - Eastern Connecticut Hematology/Oncology Assoc., Norwich, Connecticut
  - Cancer Specialists, LLC - Department of Clinical Research, Jacksonville, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital - Clinical Research, Decatur, Illinois
  - Baptist Health Lexington Oncology Associates, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Medical Center, Detroit, Michigan
  - Health Midwest Ventures Group, Inc d/b/a HCA MidAmerica Division, LLC - Menorah Medical Center - Oncology Account, Kansas City, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology, P.A. - Sugarland, Sugar Land, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Argentina (6):
  - Centro de Oncologia e Investigacion Buenos Aires, Berazategui
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Instituto de Oncología de Rosario, Rosario
  - Centro Medico San Roque S.R.L., San Miguel de Tucumán
- Belgium (4):
  - Universitair Ziekenhuis Brussel - Geriatrie, Brussels
  - Jessa Ziekenhuis Hospital, Hasselt
  - UZ Leuven, Pellenberg
  - CHU Mont-Godinne, Yvoir
- Brazil (6):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza
  - Hospital São Lucas da PUCRS, Porto Alegre
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - NOB - Núcleo de Oncologia da Bahia, Salvador
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia - Faculdade de Medicina do ABC, Santo André
- Canada (3):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Tom Baker Cancer Centre, Alberta
  - Stronach Regional Cancer Centre - at Southlake, Ontario
- China (3):
  - Peking University Cancer Hospital, Beijing
  - Guangdong General Hospital, Guangzhou
  - Shanghai Cancer Hospital, Fudan University, Shanghai
- France (7):
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Maison du Ha, Pessac, Gironde
  - Centre Hospitalier Intercommunal de Créteil - Service de Pneumologie, Créteil, Val De Marne
  - Hôpital Nord - AP-HM Marseille# - Service d'Oncologie Multidisciplinaire, Bouches-du-Rhône
  - Centre Léon Bérard, Lyon
  - CHU Rennes - Hopital Pontchaillou - service de pneumologie, Rennes
  - ICO - Site René Gauducheau, Saint-Herblain
  - CHU de Toulouse - Hôpital Larrey - Service de Pneumologie et Oncologie Pneumologique, Toulouse
- Germany (6):
  - Vivantes Klinikum Am Urban - Haematologie und Onkologie, Berlin
  - Asklepios Fachkliniken Muenchen-Gauting - Abteilung Internistische Onkologie, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Medizinische Hochschule Hannover - Pneumologie, Hanover
  - Universitaetsklinikum Schleswig- Holstein Campus Luebeck, Lübeck
  - Universitaetsklinikum Regensburg - Klinik und Poliklinik fuer Innere Medizin II, Regensburg
- Greece (4):
  - 251 General Air Force Hospital, Athens
  - General Hospital of Athens of Chest Disease "SOTIRIA", Athens
  - University General Hospital of Heraklion "PAGNI", Heraklion
  - General Hospital Papageorgiou-2nd Department of Dermatalogy, Thessaloniki
- Hong Kong (3):
  - Princess Margaret Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong - Emergency Medicine, Shatin
- Italy (7):
  - Azienda Ospedaliera San Giuseppe Moscati - U.O Oncologia Medica, Avellino
  - IRCCS Centro di Riferimento Oncologico - Oncologia Medica A, Aviano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi - Oncologia Medica, Bologna
  - Azienda Ospedaliera Univ. Policlinico Gaspare Rodolico - Unità Operativa di Oncologia, Catania
  - Azienda Ospedaliero Universitaria Mater Domini-Campus Universitario - Centro Oncologico, Catanzaro
  - Fondazione IRCCS Istituto Nazionale dei Tumori - Medicina Oncologica I, Milan
  - Università degli studi della Campania Luigi Vanvitelli - Dipartimento di Oncologia, Napoli
- Japan (8):
  - NHO Hokkaido Cancer Center - Dept of Respiratory Medicine, Sapporo, Hokkaido
  - National Cancer Center Hospital - Dept of Respiratory Medicine, Chūōku
  - Saitama Medical University International Medical Center - Dept of Respiratory Medicine, Hidaka-shi
  - Saitama Cancer Center, Kitaadachigun
  - Cancer Institute Hospital of JFCR - Dept of Respiratory Medicine, Kōtoku
  - Kurume University Hospital, Kurume-shi
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Kindai University Hospital, Osakasayama-sh
- Netherlands (6):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG) - Parent, Groningen
  - Maastricht University Medical Center - Dept of Medical Oncology, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - St. Elisabeth Ziekenhuis - Parent, Tilburg
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital del Mar - Servicio de Oncologia, Barcelona
  - Hospital Universitari Quiron Dexeus - Servicio de Oncologia Medica, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena - Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio - Servicio de Oncologia, Seville
  - Hospital Universitari i Politecnic La Fe - Servicio de Oncologia Medica, Valencia
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Adana Numune Training and Research Hospital - Cardiology Department, Adana
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital - Oncology Department, Ankara
  - Trakya University Medical Faculty - Medical Oncology, Edirne
  - Kocaeli University Research and Application Hospital, Kocaeli
- Ukraine (6):
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU - Ch of Oncology and MR, Dnipro
  - CI Transcarpathian Cl Onc Center Dep of Surgery#1 SHEI Ivano-Frankivsk NMU - Chair of Oncology, Ivano-Frankivsk
  - Communal Non-profit Enterprise Regional Center of Oncology - Parent, Kharkiv
  - Medical and Preventive Treatment Institution Volyn Regional Oncological Dispensary - Dept of Oncochemotherapy, Lutsk
  - CCCH City Oncological Center SHEI Uzhgorod NU - Ch of R&O of Faculty of PGE&PUT, Uzhhorod
  - Medical center "Oncolife", Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Brown T, Pilkington G, Bagust A, Boland A, Oyee J, Tudur-Smith C, Blundell M, Lai M, Martin Saborido C, Greenhalgh J, Dundar Y, Dickson R. Clinical effectiveness and cost-effectiveness of first-line chemotherapy for adult patients with locally advanced or metastatic non-small cell lung cancer: a systematic review and economic evaluation. Health Technol Assess. 2013 Jul;17(31):1-278. doi: 10.3310/hta17310. PMID 23886301
- [Result] Cho BC, Lee JS, Wu YL, Cicin I, Dols MC, Ahn MJ, Cuppens K, Veillon R, Nadal E, Dias JM, Martin C, Reck M, Garon EB, Felip E, Paz-Ares L, Mornex F, Vokes EE, Adjei AA, Robinson C, Sato M, Vugmeyster Y, Machl A, Audhuy F, Chaudhary S, Barlesi F. Bintrafusp Alfa Versus Pembrolizumab in Patients With Treatment-Naive, Programmed Death-Ligand 1-High Advanced NSCLC: A Randomized, Open-Label, Phase 3 Trial. J Thorac Oncol. 2023 Dec;18(12):1731-1742. doi: 10.1016/j.jtho.2023.08.018. Epub 2023 Aug 18. PMID 37597750
- [Derived] Milenkovic-Grisic AM, Terranova N, Mould DR, Vugmeyster Y, Mrowiec T, Machl A, Girard P, Venkatakrishnan K, Khandelwal A. Tumor growth inhibition modeling in patients with second line biliary tract cancer and first line non-small cell lung cancer based on bintrafusp alfa trials. CPT Pharmacometrics Syst Pharmacol. 2024 Jan;13(1):143-153. doi: 10.1002/psp4.13068. Epub 2023 Dec 13. PMID 38087967
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0037
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Participants received intravenous infusion of Pembrolizumab at a dose of 200 milligrams (mg) once every 3 weeks until confirmed progression of disease, death, unacceptable toxicity, or study withdrawal.
Period: Overall Study
Arm/Group | M7824 | Pembrolizumab
Started | 152 | 152
Treated | 151 | 152
Completed | 151 | 152
Not Completed | 1 | 0
Not completed — Randomized, not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomized to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | M7824 | Pembrolizumab | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (9.56) | 67 (10.17) | 67 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 36 | 78
  Male | 110 | 116 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 138 | 138 | 276
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 55 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 91 | 79 | 170
  Unknown or Not Reported | 7 | 14 | 21
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Independent Review Committee (IRC)
Description: Progression free survival was defined as the time from randomization of study intervention until the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from randomization of study drug until the first documentation of PD or death, assessed approximately up to 746 days
Population: Full analysis set included all participants who were randomized to study intervention.
Measure: Median (Full Range); unit: months
Arm/Group | M7824 | Pembrolizumab
Number analyzed (Participants) | 152 | 152
months | 7.0 [0.0 to 19.4] | 11.1 [0.0 to 18.0]

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization of study intervention to the date of death due to any cause. The overall survival was analyzed by using the Kaplan-Meier method.
Time Frame: Time from randomization of study drug assessed approximately up to 843 days
Population: Full analysis set included all participants who were randomized to study intervention.
Measure: Median (Full Range); unit: months
Arm/Group | M7824 | Pembrolizumab
Number analyzed (Participants) | 152 | 152
months | 21.1 [0.2 to 22.1] | 22.1 [0.1 to 26.4]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on treatment period. TEAEs included serious AEs and non-serious AEs. Treatment-related TEAEs: reasonably related to the study intervention.
Time Frame: Time from first treatment assessed up to approximately 843 days
Population: Safety analysis set included all participants who were administered at least one dose of M7824 or Pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | M7824 | Pembrolizumab
Number analyzed (Participants) | 151 | 152
Participants
  Participants with any TEAE | 150 | 145
  Participants with any serious TEAE | 90 | 61
  Participants with any Treatment Related TEAEs | 124 | 105

4. Secondary Outcome: Percentage of Participants With Unconfirmed Best Overall Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: Percentage of participants with unconfirmed best overall response that is at least one overall assessment of complete response (CR) or partial response (PR) reported here.
Time Frame: as for outcome 1
Population: Full analysis set included all participants who were randomized to study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824 | Pembrolizumab
Number analyzed (Participants) | 152 | 152
percentage of participants | 46.7 [38.6 to 55.0] | 51.3 [43.1 to 59.5]

5. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: DOR was defined for participants with objective response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC. Results were calculated based on Kaplan-Meier estimates.
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 746 days
Population: Full analysis set included all participants who were randomized to study intervention. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824 | Pembrolizumab
Number analyzed (Participants) | 71 | 78
months | NA [NA to NA] — Due to small number of events, estimates (Median, lower limit and upper limit) from Kaplan-Meier survival curves could not derive. | NA [13.5 to NA] — Due to small number of events, estimates (Median and upper limit) from Kaplan-Meier survival curves could not derive.

ADVERSE EVENTS:
Time Frame: Time from first treatment assessed up to approximately 843 days
Description: Safety analysis set included all participants who were administered at least one dose of M7824 or Pembrolizumab.
Arm/Group | M7824 | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 49/151 | 43/152
Serious Adverse Events (participants affected / at risk) | 90/151 | 61/152
Other Adverse Events (participants affected / at risk) | 140/151 | 135/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M7824 (N=151) | Pembrolizumab (N=152)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Death (General disorders) | 1 | 1
Disease progression (General disorders) | 6 | 7
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Hyperthermia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 12
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 2
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Keratoacanthom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M7824 (N=151) | Pembrolizumab (N=152)
Anaemia (Blood and lymphatic system disorders) | 46 | 18
Hyperthyroidism (Endocrine disorders) | 6 | 10
Hypothyroidism (Endocrine disorders) | 17 | 23
Abdominal pain upper (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 16 | 22
Diarrhoea (Gastrointestinal disorders) | 24 | 24
Dyspepsia (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 19 | 20
Vomiting (Gastrointestinal disorders) | 14 | 10
Asthenia (General disorders) | 26 | 30
Chest pain (General disorders) | 8 | 6
Fatigue (General disorders) | 30 | 26
Oedema peripheral (General disorders) | 14 | 13
Pyrexia (General disorders) | 28 | 15
Pneumonia (Infections and infestations) | 8 | 21
Upper respiratory tract infection (Infections and infestations) | 9 | 2
Urinary tract infection (Infections and infestations) | 11 | 4
Alanine aminotransferase increased (Investigations) | 19 | 16
Amylase increased (Investigations) | 9 | 9
Aspartate aminotransferase increased (Investigations) | 23 | 14
Blood alkaline phosphatase increased (Investigations) | 18 | 11
Blood bilirubin increased (Investigations) | 9 | 3
Blood creatinine increased (Investigations) | 9 | 13
Blood thyroid stimulating hormone increased (Investigations) | 2 | 8
Gamma-glutamyltransferase increased (Investigations) | 19 | 16
Lipase increased (Investigations) | 12 | 7
Weight decreased (Investigations) | 10 | 7
Decreased appetite (Metabolism and nutrition disorders) | 25 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 10
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 0
Dizziness (Nervous system disorders) | 12 | 8
Headache (Nervous system disorders) | 14 | 14
Insomnia (Psychiatric disorders) | 16 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 27 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 52 | 42
Rash (Skin and subcutaneous tissue disorders) | 48 | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 8 | 5
Hypertension (Vascular disorders) | 3 | 10
Hypotension (Vascular disorders) | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT03631706/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT03631706/SAP_001.pdf